CLINICAL TRIAL: NCT04683614
Title: Intraoperative Norepinephrine Versus Fresh Frozen Plasma in Patients Undergoing HIPEC to
Brief Title: Intraoperative Norepinephrine Versus Fresh Frozen Plasma in Patients Undergoing HIPEC to Reduce Renal Insult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Principal Investigator, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201920025.2P
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh frozen plasma (Experimental): early administration of fresh frozen plasma
  Interventions: Biological: Fresh frozen plasma
- Low dose norepinephrine (Experimental): low dose epinephrine 5 mic/kg/hr
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — 5 mic/kg/hr norepinephrine
  Other Names: low dose norepinephrine
  Arms: Low dose norepinephrine
Biological: Fresh frozen plasma — early administration of fresh frozen plasma
  Other Names: Blood products
  Arms: Fresh frozen plasma

SUMMARY:
comparing the effect of low dose norepinephrine infusion versus fresh frozen plasma in patients undergoing HIPEC to reduce renal insult

DETAILED DESCRIPTION:
To compare the efficacy of maintaining intraoperative hemodynamic stability through infusing low dose norepinephrine versus fresh frozen plasma in patients undergoing cytoreductive surgery and heated intraperitoneal chemotherapy in cancer patients undergoing cytoreductive surgery and heated intraperitoneal chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* World Health Performance Status ≤2
* scheduled for CRS/HIPEC operations

Exclusion Criteria:

* patient's refusal
* allergy to any of the used drugs
* impaired renal or liver functions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Renal insult | 24 hours
  Creatinine level increase 0.3 mg/dl above preoperative baseline

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt